CLINICAL TRIAL: NCT05129969
Title: SMARAGD - Clinical Research Platform on Ovarian, Fallopian Tube, Primary Peritoneal and Endometrial Cancer Treatment and Outcomes
Brief Title: Registry Platform Ovarian and Endometrial Cancer
Acronym: SMARAGD
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-110401
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Ovary Neoplasm; Endometrial Neoplasms; Carcinoma, Ovarian; Carcinoma; Neoplasm, Ovarian
Keywords: Registry; Health service research; Epidemiology; Germany; Palliative treatment; Palliative care
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ovarian cancer: Female patients with high grade OC (advanced or metastatic epithelial ovarian, fallopian tube and primary peritoneal cancer):
  * with newly diagnosed FIGO stage IIb-IV OC who are starting systemic treatment, independent of the treatment intention (adjuvant/curative or palliative) or
  * with recurrent/relapsed disease, who received any previous systemic anti-tumor treatment and who are now starting their systemic treatment for first recurrent/relapsed disease.
  Interventions: Other: Physician's choice according to patient's needs.
- Endometrial cancer: Female patients with locally advanced and inoperable or metastatic EC (FIGO stage III-IV) who are starting systemic first-line therapy.
  Interventions: Other: Physician's choice according to patient's needs.

INTERVENTIONS:
Other: Physician's choice according to patient's needs. — Routine care as per site standard.

SUMMARY:
The purpose of the project is to set up a national, prospective, longitudinal, multicenter cohort study, a tumor registry platform, to document uniform data on characteristics, molecular diagnostics, treatment and course of disease, to collect patient-reported outcomes and to establish a decentralized biobank for patients with advanced or metastatic ovarian cancer (OC) or advanced or metastatic endometrial cancer (EC) in Germany.

DETAILED DESCRIPTION:
SMARAGD is a national, prospective, open-label, longitudinal, non-interventional multicenter cohort study (tumour registry platform) to describe treatment in routine clinical practice of ovarian, fallopian tube, primary peritoneal and endometrial patients in routine care in Germany.

The registry will follow patients for up to three years with the aim to identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented.

Health-related quality of life (HRQoL) will be evaluated for up to three years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed high grade OC (advanced or metastatic epithelial ovarian, fallopian tube and primary peritoneal cancer):

  * patients with FIGO stage IIb-IV OC who are starting systemic treatment or
  * patients with recurrent/relapsed disease, who received any previous systemic anti-tumor treatment and who are now starting systemic treatment for recurrent/relapsed disease.
* Locally advanced and inoperable or metastatic EC (FIGO stage III-IV) who are starting systemic first-line therapy.
* Signed and dated informed consent (IC):

  * Patients participating in PRO module: IC before first therapy cycle
  * Patients not participating in PRO module: IC no later than six weeks after start of first therapy cycle

Exclusion Criteria:

* newly diagnosed early-stage OC (FIGO stage I-IIa)
* Low grade mOC OR
* Early-stage EC (FIGO stage I-II)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian or endometrial cancer.
Study Population: Adult female patients with (metastatic) ovarian cancer (FIGO stage IIb-IV) or (metastatic) endometrial cancer (FIGO stage III-IV) starting systemic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1975 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Course of treatment (treatment reality). | 3 years per patient
  Documentation of anamnestic data and therapy sequences.

SECONDARY OUTCOMES:
Best Response. | 3 years per patient
  Documentation of response rates per line of treatment.
Progression-free survival. | 3 years per patient
  Documentation of progression-free survival per line of treatment.
Overall survival. | 3 years per patient
  Documentation of overall survival per line of treatment.
Health-related quality of life (Patient-reported outcome, PRO). | 3 years per patient
  Functional Assessment of Cancer Therapy - Ovarian (FACT-O), a 39 item questionnaire covering Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being and Ovarian Cancer Subscale
Health-related quality of life (Patient-reported outcome, PRO). | 3 years per patient
  Functional Assessment of Cancer Therapy - Endometrial (FACT-En), a 43 item questionnaire covering Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being and Endometrial Cancer Subscale

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Decker, Prof.Dr., Study Chair — Ravensburg; Ingolf Juhasz-Böss, Prof.Dr., Study Chair — Freiburg; Elmar Stickeler, Prof.Dr., Study Chair — Aachen; Dirk Watermann, Prof.Dr., Study Chair — Freiburg; Anja Welt, Dr., Study Chair — Essen; Achim Wöckel, Prof.Dr., Study Chair — Würzburg
Locations (1):
- Multiple sites all over Germany, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No